CLINICAL TRIAL: NCT01689636
Title: CLINICAL STUDY OF A SINGLE-CENTER CLINICAL STUDY TO EVALUATE THE SAFETY AND BIODISTRIBUTION OF TECHNETIUM Tc 99m EC20 IN NORMAL VOLUNTEERS AND OVARIAN CANCER PATIENTS
Brief Title: Safety and Biodistribution of Technetium Tc 99m EC20 in Normal Volunteers and Ovarian Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.1
Record Dates: First submitted 2012-09-09; First posted 2012-09-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Healthy Volunteers
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

ARMS (1):
- Single-center, open-label (Experimental): The study was designed as a single-center, open-label clinical study to evaluate the safety, pharmacokinetics, dosimetry and metabolism of Tc 99m EC20 in normal volunteers and in patients with known or suspected ovarian cancer.
  Eight subjects were to be enrolled at one center: four normal subjects, four patients with ovarian cancer. Each subject was to receive a single injection of Tc 99m EC20 complex composed of 0.1 mg ligand (EC20) and 15 - 20 mCi of Tc 99m. Two (2) of the 4 normal subjects and 2 of the 4 patients were to receive an injection of 0.25-2.0 mg folic acid 1-2 minutes prior to the injection of Tc 99m EC20.
  Interventions: Drug: Tc 99m EC20

INTERVENTIONS:
Drug: Tc 99m EC20

SUMMARY:
Open-label, single-center, single-treatment group, baseline-controlled (for safety) study of the safety and biodistribution of Technetium Tc 99m EC20 in four normal subjects and four subjects with known or suspected ovarian cancer.

DETAILED DESCRIPTION:
This was a single-center, open-label evaluation of a single injection of Tc 99m EC20 containing 0.1 mg EC20 labeled with 15 - 20 mCi of technetium-99m in normal volunteers and patients with known or suspected ovarian cancer. Two normal volunteers and two patients also were to receive an injection of 0.25 - 2.0 mg folic acid 1 to 2 minutes prior to the injection of Tc 99m EC20. Serial blood samples and urine were collected during the 24-hour period following each injection for pharmacokinetic evaluation. Serial whole body images were acquired during the 24-hour postdose period for dosimetry evaluations. Safety was monitored through predose and postdose physical examinations, electrocardiograms (ECGs), vital signs and clinical laboratory evaluations. Adverse events were monitored from the time of signing of Informed Consent to 24 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were to be females 18 years of age or older who met the following criteria:

  1. The four normal subjects were to be normal, as established by medical history, physical examination, and laboratory data, including CBC, serum chemistry, and urinalysis.
  2. The two subjects with obvious advanced stage ovarian cancer were to have either histopathologically proven stage 3 or 4 disease or clinically obvious disease defined by 2 of the following 3 conditions: (1) pelvic mass (2) omental "caking", or (3) ascites.
  3. Subjects were to have newly diagnosed, treatment refractory, or recurrent disease. Subjects were to be treatment naïve or at least 2 months since last non-surgical treatment. Subjects were to have normal kidney and liver function.
  4. The two subjects with suspected ovarian cancer were to have a known mass. Subjects were to have normal kidney and liver function.
  5. Subjects were to provide informed consent prior to enrollment.

Exclusion Criteria:

* The following subjects were to be excluded:

  1. Subject was pregnant or breast-feeding.
  2. Subject was simultaneously participating in another investigative drug or device study, or had completed follow-up phase of any previous study within 30 days prior to enrollment in this study.
  3. Subject had a known history of chronic abuse of drugs or alcohol or had tested positive in the pre-study urine drug abuse screen.
  4. Subject was currently taking folic acid supplements and could not stop taking the supplements for a period of 3 days (2 days prior to the study and one day after last imaging procedure).
  5. Subject had physical condition that was unsuitable for radionuclide imaging.
  6. Subject had been administered another radiopharmaceutical that would interfere with the assessment of the biodistribution of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2000-08; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Determine the biodistribution and excretion of the radioactive drug substance (Technetium Tc 99m EC20) and estimate the radiation absorbed dose | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States